CLINICAL TRIAL: NCT02302521
Title: Examining the Clinical Utility of Motion Immune MRI Across Multiple Patient Populations
Brief Title: Motion Immune Magnetic Resonance Imaging (MRI)
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00057343
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2016-07

CONDITIONS: Parkinson's Disease
Keywords: MRI
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (4):
- Healthy Younger Adults: Age: 20-30. Gender: male or female. No neurological conditions.
  Interventions: Device: Multiplex Sensitivity Encoding (MUSE)
- Healthy Older Adults: Age: 50-70. Gender: male or female. No neurological conditions.
  Interventions: Device: Multiplex Sensitivity Encoding (MUSE)
- Parkinson's disease: Gender: male or female. Tremor dominant Parkinson's disease.
  Interventions: Device: Multiplex Sensitivity Encoding (MUSE)
- Healthy Children: Age: 4-8. Gender:male or female. No neurological conditions.
  Interventions: Device: Multiplex Sensitivity Encoding (MUSE)

INTERVENTIONS:
Device: Multiplex Sensitivity Encoding (MUSE) — It is an algorithm for MRI post-processing/image reconstruction (see reference: Chen).

SUMMARY:
The purpose of this study is to evaluate our recently developed MRI reconstruction strategy for producing artifact-free neuro and abdominal MRI data. The new reconstruction strategies, including 1) REKAM and 2) MUSE, are capable of effectively removing motion-related artifacts resulting from global and local motion during neuro and free-breathing abdominal MRI scans, without modifying the MRI pulse sequences and protocols that are currently used in clinical scans. The study team aims to recruit 60 subjects across multiple challenge patient populations: 10 healthy young adults (age 20-30) and 10 healthy older adults (aged 50-70) for abdominal MRI, as well as 20 tremor dominant PD patients and 20 children (age 4-8) for brain MRI scans. There are no known risks in taking MRIs and a unique code will be assigned to each participant to protect their PHI.

ELIGIBILITY:
Inclusion Criteria:

1. subject's age is within one of the following age ranges (4-8, 20-30, or 50-70 years old);
2. male or female;
3. healthy volunteer or diagnosed with PD ; and
4. devoid of the following exclusion criteria.

Exclusion Criteria:

1. claustrophobia or other MRI contraindications (including pregnancy);
2. diagnosis for dementia (Alzheimer's, Lewy Body, or Vascular);
3. symptomatic psychotic disorders;
4. depression with psychotic symptoms;
5. other psychotic or schizophrenic disorders;
6. recent neuroleptic treatment;
7. history of cardiovascular disease;
8. history of stroke or Transient Ischemic Attack;
9. cancer (other than skin cancer) within the last three years;
10. hospitalization for neurological/psychiatric condition;
11. significant handicaps (e.g., visual or hearing loss, mental retardation) that would interfere with neuropsychological testing or the ability to follow study procedures; or
12. any other factor that in the investigators' judgment may affect patient safety or compliance.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: There are 4 separate cohorts of patients. Please see earlier section. 60 subjects will participate in our study.
  * 10 healthy younger adult volunteers (ages 20 to 30)
  * 10 healthy older adult volunteers (ages 50 to 70) will be recruited for
  * 20 tremor-dominant patients with clinically diagnosed Parkinson's disease
  * 20 healthy children (4 to 8 y.o.)
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2016-11-26 (Actual); Study Completion 2016-11-26 (Actual)

PRIMARY OUTCOMES:
Rating of image quality (based on 8 criteria) by multiple radiologists (blind to reconstruction method) | 1 day (At time of image analysis)
  The ratings will be compared to compare the quality of images processed with MUSE versus conventional reconstruction methods

CONTACTS AND LOCATIONS:
Overall Officials: Nan-kuei Chen, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Chen NK, Guidon A, Chang HC, Song AW. A robust multi-shot scan strategy for high-resolution diffusion weighted MRI enabled by multiplexed sensitivity-encoding (MUSE). Neuroimage. 2013 May 15;72:41-7. doi: 10.1016/j.neuroimage.2013.01.038. Epub 2013 Jan 28. PMID 23370063